CLINICAL TRIAL: NCT04210492
Title: Phase IB/II Trial Of Dose-Deescalated 3-Fraction Stereotactic Body Radiotherapy For Centrally Located Lung Cancer
Brief Title: Dose-Deescalated 3-Fraction Stereotactic Body Radiotherapy For Centrally Located Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000025868
Record Dates: First submitted 2019-12-10; First posted 2019-12-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: The intervention group will be compared with historical controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 45 Gy (Experimental): Deescalated 3-fraction stereotactic body radiotherapy regimen to 45 Gy in 3 fractions.
  Interventions: Radiation: 45 Gray (Gy) regimen

INTERVENTIONS:
Radiation: 45 Gray (Gy) regimen — Deescalated 3-fraction stereotactic body radiotherapy regimen to 45 Gy in 3 fractions.

SUMMARY:
The purpose of this trial is to test a deescalated 3-fraction stereotactic body radiotherapy (SBRT) regimen to 45 Gray (Gy) in 3 fractions for centrally located thoracic tumors.

DETAILED DESCRIPTION:
The purpose of this trial is to test a deescalated 3-fraction SBRT regimen to 45 Gy in 3 fractions for centrally located thoracic tumors in a phase II trial. This will provide prospectively collected data on the safety and efficacy of a three-fraction regimen in the previously defined "No Fly Zone" for both primary non-small cell lung cancer (NSCLC) and for lung metastases of any histology. This registration describes the design and eligibility criteria for the 36 NSCLC subjects the investigators plan to enroll. Local control, cancer-specific survival, and overall survival results from the NSCLC patients will be compared to both 3- and 5-fraction historical controls, specifically RTOG 0236 and 0813 results.

The outcomes of the metastatic patients will also be reported.

There will also be a quality-of-life component to the study to assess the impact of a shorter overall treatment time and the clinical impact of radiation side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Lung tumors will be ≤ 5 cm and centrally located, meaning any portion of gross tumor volume located within 2 cm of (but not abutting) the proximal bronchial tree (trachea, carina, right and left main bronchi, right and left upper lobe bronchi, bronchus intermedius, right middle lobe bronchus, lingular bronchus, right and left lower lobe bronchi), or within 2 cm of (whether abutting or not) major vessels, esophagus, or heart (based on RTOG and MD Anderson Cancer Center definitions 33,34). Multiple concurrent isocenters are allowed if at least one tumor meets the above criteria, and if all dose constraints for the plan summation can be met. These concurrent tumors other than study target lesion can be treated as per SOC and does not necessarily have to meet the above size limit. The PI will review and prospectively approve any lesions abutting these organs.
2. ECOG Performance Status of 0-2
3. Age > 18
4. Patients must sign a study-specific consent form.

Exclusion Criteria:

1. Prior history of radiotherapy near target lesion resulting in overlapping treatment fields. Previously irradiated will be defined as OAR structures receiving the following doses (in <3Gy per fraction):

   * Spinal cord previously irradiated to > 40 Gy
   * Brachial plexus previously irradiated to > 50 Gy
   * Small intestine, large intestine, or stomach previously irradiated to > 45Gy
   * Brainstem previously irradiated to > 50 Gy
   * Lung previously irradiated with prior V20Gy > 35%
2. Active systemic, pulmonary, or pericardial infection
3. Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
4. Pregnant or lactating
5. Any other medical condition or reason that, in the opinion of the investigator, would preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Safety of the stereotactic body radiotherapy regimen (SBRT) | From administration of SBRT up to 2 years post-SBRT
  Safety will be assessed by acute (defined as within 90 days of stereotactic body radiotherapy (SBRT)) and late (from 91 days through 2 years post-SBRT) toxicities. Toxicities are based on (Common Terminology Criteria for adverse events) CTCAE v. 5 criteria
local control (LC) of 3-fraction stereotactic body radiotherapy | Up to 10 years post-enrollment.
  The absence of primary tumor failure. Primary tumor failure is defined as Increase in tumor dimension of 20%.

SECONDARY OUTCOMES:
lobar control | Up to 10 years post-enrollment.
  Absence of primary tumor failure or involved lobe failure or both.
regional control | Up to 10 years post-enrollment.
  Absence of measurable tumor within lymph nodes along the natural lymphatic drainage typical for the location of the treated primary disease only with dimension of at least 1.0 cm on imaging studies (preferably computer tomography scans) within the lung, bronchial hilum, or the mediastinum.
distant control | Up to 10 years post-enrollment.
overall survival | Up to 10 years post-enrollment.
progression-free survival | Up to 10 years post-enrollment.

OTHER OUTCOMES:
organ at risk (OAR) dosimetry | Up to 10 years post-enrollment.
quality of life (QOL) | baseline and up to 5 years.
  QOL will be measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). Each item of this 30-item questionnaire is measured on a scale ranging from 1-4, with higher scores signaling lower quality of life. The total possible score is 120. Quality of life will be measured longitudinally, as one outcome. This outcome will be measured at baseline, on the last day of treatment and at 1, 4, 8, and 12 months post-treatment. Thereafter, quality of life will be measured every 6 months, up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Park, MD, MPH, Principal Investigator — Yale University
Locations (6):
- United States (6):
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital - Hamden Care Center, Hamden, Connecticut
  - Smilow Cancer Hospital, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center - Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut

IPD SHARING:
Plan to Share IPD: No